CLINICAL TRIAL: NCT01367548
Title: A Phase II Double-Blind Randomized Parallel Group Study of Intravenous (IV) Methylnaltrexone (MNTX) in the Prevention of Post-Operative Ileus
Brief Title: Intravenous (IV) Methylnaltrexone (MNTX) in the Prevention of Post-Operative Ileus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Tage Ramakrishna, MD, Progenics Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNTX 203
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: IV Methylnaltrexone (MNTX)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Methylnaltrexone (MNTX)
  Arms: Arm 1
Drug: Placebo
  Arms: Arm 2

SUMMARY:
A double-blind, randomized, parallel-group study designed to evaluate the safety and activity of IV MNTX in the treatment of Post-Operative Ileus (POI) in patients who underwent segmental colectomies via laparotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 yrs or older
2. Patients who have undergone a segmental colectomy
3. Must be receiving opioids via IV.

Exclusion Criteria:

1. Patients who received any experimental drug in the last 30 days
2. Patients receiving spinal medication for post-operative pain relief
3. Patients who have undergone operations for complications related to inflammatory bowel disease
4. Patients with recent history of abdominal radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-07; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Time to tolerance of liquids | 7 days
  To assess the activity of parenterally administered MNTX compared with placebo in shortening the duration of or preventing post-operative ileus in patients who have undergone segmental colectomies.

SECONDARY OUTCOMES:
Time to first bowel movement | 7 days
  To assess the activity of parenterally administered MNTX compared with placebo in shortening the duration of or preventing post-operative ileus in patients who have undergone segmental colectomies.
Time to tolerance of solid foods | 7 days
  To assess the activity of parenterally administered MNTX compared with placebo in shortening the duration of or preventing post-operative ileus in patients who have undergone segmental colectomies.
Time to first micturition post foley catheter removal | 7 days
  To assess the activity of parenterally administered MNTX compared with placebo in shortening the duration of or preventing post-operative ileus in patients who have undergone segmental colectomies.
Time to hospital discharge | 7 days
  To assess the activity of parenterally administered MNTX compared with placebo in shortening the duration of or preventing post-operative ileus in patients who have undergone segmental colectomies.

CONTACTS AND LOCATIONS:
Overall Officials: Tage Ramakrishna, MD, Study Director — Progenics Pharmaceuticals, Inc.
Locations (1):
- Progenics Pharmaceuticals, Inc., Tarrytown, New York, United States